CLINICAL TRIAL: NCT01764542
Title: Critical Assessment of Routine Surveillance of Asymptomatic Patients With Ulcerative Colitis With Ileal Pouch-anal Anastomosis and Risk Factors for Dysplasia - is There a Rationale?
Brief Title: Development of Dysplasia in the Pelvic Pouch in Patients With Ulcerative Colitis (UC) and Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mattias Block (Other)
Responsible Party: Sponsor-Investigator, Mattias Block, Doctor, Surgeon, MD, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GLS-249941
Record Dates: First submitted 2012-09-27; First posted 2013-01-09 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Ulcerative Colitis; Dysplasia; Surgery
Keywords: Ulcerative colitis; dysplasia; risk factor; surgery
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Endoscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopy and biopsy (Other): Endoscopy with biopsy taken Endoscopy and biopsy Blood samples Questionnaire
  Interventions: Procedure: Endoscopy and biopsy

INTERVENTIONS:
Procedure: Endoscopy and biopsy — Endoscopy with biopsy of the ileo-anal pouch and the ileo-anal anastomosis Blood samples

SUMMARY:
The purpose of this study is to study development of dysplasia in the ileal mucosa among patients with Ulcerative Colitis and who previous have hade risk factors for developing cellular changes/dysplasia, i.e. previous dysplasia and/or carcinoma in their specimen.

DETAILED DESCRIPTION:
Objective Some of the rare complications reported in patients with an ileal pouch-anal anastomosis (IPAA) after colectomy for chronic ulcerative colitis are dysplasia and carcinoma. The supposed pathway is for the ileal pouch mucosa to go through adaptational changes then to progress through the phases of chronic pouchitis, dysplasia and subsequently to adenocarcinoma. The purpose of this study is to study development of dysplasia in the ileal mucosa among patients with Ulcerative Colitis and who previous have hade risk factors for developing cellular changes/dysplasia, i.e. previous dysplasia and/or carcinoma in their specimen.

Methods In a cohort of 680 patients having IPAA with a median follow-up time of 18 years, 75 patients with risk factors for dysplasia were identified. Sixty-five patients were eligible for inclusion, fifty-six patients accepted to participate in the study. Patients are invited for clinical examination, endoscopy with macroscopic evaluation as well as mucosal biopsies. The biopsies are reviewed and evaluated by two independent pathologists, experienced in colonic pathology, concerning morphological changes, dysplasia and potential carcinoma Results Architectural structural changes, inflammation and reactive atypia is noted in the rectal cuff and ileal pouch. So far, none of the biopsies showed genuine dysplasia after a follow up for 18 years (Range 12-23 years). In this respect there is full agreement between the two pathologists.

Further microscopic evaluation are planned for the rest of the participating patients.

ELIGIBILITY:
Inclusion Criteria:

* UC (Ulcerative Colitis)
* IPAA
* risk factor for dysplasia

Exclusion Criteria:

* Not able to give consent
* CD (Crohns disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Presence of dysplasia in patients with Ulcerative Colitis and Ileal Pouch-Anal Anastomosis | Up to 7 days
  The study ends at above mentioned date. After that, microscopic evaluation, statistics and analysis will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Börjesson, Surgeon, Study Chair — Department of Surgery, Sahlgrenska, Göteborg
Locations (1):
- Department of Surgery, Inst for Clinical Sciences, Sahlgrenska University Hospital, Gothenburg, Göteborg, Sweden